CLINICAL TRIAL: NCT01222676
Title: A Phase II Study of Neoadjuvant Cisplatin and Gemcitabine Plus Sorafenib for Patients With Transitional-Cell Carcinoma of the Bladder
Brief Title: Cisplatin, Gemcitabine Hydrochloride, and Sorafenib Tosylate in Treating Patients With Transitional Cell Cancer of the Bladder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ITA-MIL-IRCCS-INT-52/10; CDR0000686602 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2010-022653-41; EU-21077
Record Dates: First submitted 2010-10-15; First posted 2010-10-18 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2010-10

CONDITIONS: Bladder Cancer
Keywords: transitional cell carcinoma of the bladder; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Sorafenib; Neoadjuvant Therapy; Fluorodeoxyglucose F18

INTERVENTIONS:
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: sorafenib tosylate
Other: imaging biomarker analysis
Other: laboratory biomarker analysis
Procedure: computed tomography
Procedure: neoadjuvant therapy
Radiation: fludeoxyglucose F 18

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cisplatin and gemcitabine hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Sorafenib tosylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth or by blocking blood flow to the tumor. Giving cisplatin and gemcitabine hydrochloride together with sorafenib tosylate may kill more tumor cells. Giving them before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving cisplatin and gemcitabine hydrochloride together with sorafenib tosylate works in treating patients with node-negative transitional cell cancer of the bladder.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the activity (pathological complete response) of neoadjuvant cisplatin and gemcitabine hydrochloride in combination with sorafenib tosylate in patients with muscle-invasive, node-negative transitional cell carcinoma of the bladder.

Secondary

* To evaluate the safety and tolerability of this regimen in these patients.
* To determine the potential biological correlates of disease response and drug activity in tumor tissue samples before and after treatment.
* To evaluate the correlation between fludeoxyglucose F 18 positron emission tomography (18FDG-PET) and standard computed tomography (CT) results and the ability of changes of 18FDG-PET (as measured by EORTC criteria for response) to predict subsequent favorable response to treatment (pathological complete response rate and progression-free survival).

OUTLINE: Patients receive cisplatin IV over 20-30 minutes on day 1 and gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. Patients also receive sorafenib tosylate twice daily on days 1-21. starting on day 1and continuing up to Treatment repeats every 21 days for 2 courses. Patients are reassessed after course 2, those who experience disease progression or deemed unresectable are off study. Other patients continue the treatment for 2 more courses*.

NOTE: *Sorafenib tosylate are stopped 14 days prior to planned cystectomy.

No more than 30 days after completion of neoadjuvant therapy, patients undergo planned radical cystectomy with pelvic lymph-node dissection off study.

Tumor tissue and serum samples may be collected during study for additional biological studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed transitional cell carcinoma (TCC) of the bladder at the time of diagnostic transurethral resection of the bladder tumor (TURB)*

  * Muscle-invasive (T ≥ 2) disease at TURB OR clinical stage T3 or T4 disease (e.g., T2 patients will not be eligible without a histological documentation of invasive disease)
* NOTE: *Confirmation of TCC histology based on pathologic review at Fondazione Istituto Nazionale dei Tumori Milan will be required in all cases.
* Clinically node-negative (cN0) disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 2,000/µL
* ANC ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* Serum creatinine ≤ 1.5 mg/dL
* AST/ALT < 2.5 times upper limit of normal (ULN) (< 5 times ULN if due to hepatic metastases)
* Total bilirubin < 1.5 times ULN
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* Negative serology for the following infectious diseases:

  * HIV type 1 or 2
  * Hepatitis B surface antigen (active carriers)
  * Hepatitis C

PRIOR CONCURRENT THERAPY:

* No prior systemic therapies except for intravesical therapy for superficial disease
* No prior sorafenib tosylate
* No prior systemic chemotherapy
* At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response

SECONDARY OUTCOMES:
Safety and tolerability
Potential biological correlates of disease response and drug activity in tumor tissue samples before and after therapy
Correlation between 18FDG-PET and standard CT results

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Salvioni, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione Istituto Nazionale dei Tumori, Milan, Italy

REFERENCES:
- [Derived] Necchi A, Lo Vullo S, Raggi D, Perrone F, Giannatempo P, Calareso G, Togliardi E, Nicolai N, Piva L, Biasoni D, Catanzaro M, Torelli T, Stagni S, Colecchia M, Busico A, Pennati M, Zaffaroni N, Mariani L, Salvioni R. Neoadjuvant sorafenib, gemcitabine, and cisplatin administration preceding cystectomy in patients with muscle-invasive urothelial bladder carcinoma: An open-label, single-arm, single-center, phase 2 study. Urol Oncol. 2018 Jan;36(1):8.e1-8.e8. doi: 10.1016/j.urolonc.2017.08.020. Epub 2017 Sep 12. PMID 28911922